CLINICAL TRIAL: NCT06852378
Title: Comparison Between Iliopsoas Nerve Block and Femoral Nerve Block in Hip Fracture Surgeries
Brief Title: Iliopsoas Nerve Block and Femoral Nerve Block in Hip Fracture Surgeries
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hazem Khaled Abdelrazek Saeed, Assistant Lecturer of Anesthesia, Intensive Care and Pain Medicine, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: FMASU MD38/2025
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Iliopsoas Nerve Block; Femoral Nerve Block; Hip Fracture Surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Iliopsoas nerve block group: Patients will receive an Iliopsoas nerve block using 10 ml of bupivacaine 0.5%.
  Interventions: Drug: Iliopsoas nerve block
- Femoral nerve block group: Patients will receive femoral nerve block using 10 ml of bupivacaine 0.5%.
  Interventions: Drug: Femoral nerve block

INTERVENTIONS:
Drug: Iliopsoas nerve block — Patients will receive an Iliopsoas nerve block using 10 ml of bupivacaine 0.5%.
  Other Names: Bupivacaine 0.5%
  Groups: Iliopsoas nerve block group
Drug: Femoral nerve block — Patients will receive femoral nerve block using 10 ml of bupivacaine 0.5%.
  Other Names: Bupivacaine 0.5%
  Groups: Femoral nerve block group

SUMMARY:
This study aims to compare iliopsoas nerve Block (IPB) to femoral nerve block (FNB) regarding pain control, patient satisfaction, and early ambulation in patients undergoing hip fracture surgeries

DETAILED DESCRIPTION:
Hip fractures are among the most frequent fractures seen in the emergency department and orthopedic trauma teams. The terms hip fracture and neck of femur fracture are used synonymously. Both terms describe a proximal femur fracture between the femoral head and 5 cm distal to the lesser trochanter.

Iliopsoas nerve Block (IPB) is a promising motor-sparing analgesic technique that selectively targets the sensory branches of the hip joint originating from the femoral nerve and accessory obturator nerve, sparing the motor supply of quadriceps muscles.

A femoral nerve block (FNB) is a simple nerve block that can be performed easily without or under ultrasound guidance. Under ultrasound guidance, the femoral artery and femoral nerve were identified clearly, and a needle was inserted using an in-plane approach from the lateral to the medial direction. Once the needle tip's position was confirmed, 10 ml of 0.5% bupivacaine was injected adjacent to the femoral nerve.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I and II.
* Patients who are scheduled for elective surgical correction of hip fracture either through open fracture internal fixation (ORIF), partial hip arthroplasty or total hip arthroplasty.

Exclusion Criteria:

* Refusal to participate.
* Coagulopathy.
* Patients with a history of drug allergies to study drugs.
* Inability to cooperate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective, single-blind cohort study will be conducted on 80 patients scheduled for elective surgical correction of hip fracture after obtaining approval from the Research Ethical Committee of Ain Shams University. It will be conducted in the assembled operation rooms in Ain Shams University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS) score. NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed upon arrival at the post-anesthesia care unit (PACU) and at 2, 4, 6,12, 24 post-surgery.

SECONDARY OUTCOMES:
Total opioids consumption | 24 hours postoperatively
  Intravenous pethidine (25mg) will be given to be repeated after 15 min if no response up to a maximum dose of 50 mg In case of moderate to sever pain.
Assessment of quadriceps strength | 24 hours postoperatively
  The quadriceps strength will be assessed using the manual muscle testing (MMT) grade (0-5; 0: no muscle contraction, 1: muscle contraction present but unable move joint, 2: able to move joint but not resist gravity, 3: able to resist gravity but not bear substantial resistance, 4: able to resist some level of substantial resistance, 5: able to resist full resistance).
Time of ambulation | 24 hours postoperatively
  Time of ambulation will be recorded from the end of surgery till walking or moving from place to place
Patients' satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of complications | 24 hours postoperatively
  Any complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.